CLINICAL TRIAL: NCT00383058
Title: The Extract of Green Tea on Obese Women: a Randomized Double Blindness Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Taipei Hospital, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH-Greentea-06-01; NSC-95-2320-B-192-001
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Obesity
Keywords: obesity; green tea
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: the extract of green tea

SUMMARY:
The purpose of this study is to examine whether the extract of the green tea is effective on obese women.

DETAILED DESCRIPTION:
We conducted the pilot study in 2005. The initial findings showed the extract of green tea is benefit on obese women. The potential benefit include appetite lowing, lipid markers decreasing and regulating balance of obese related hormone peptides. So we designed this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-60 years old female
2. BMI>27㎞/m2
3. Signed informed consent

Exclusion Criteria:

1. Endocrine disease, e.g. thyroid disorder, pituitary disorder, and sex gland disorder.
2. Heart disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker.
3. Allergy and Immunology disease.
4. High aminotransferases ( Alanine, Aspartate >80 IU/L) or high serum Creatinine (>2.5 mg/dL)
5. Pregnant or lactating women.
6. Childbirth within 6 months.
7. Stroke or otherwise unable to exercise
8. Management for weight control within 3 months.
9. Any other conditions deemed unsuitable for trial as evaluated by the physician-in-charge.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
(Percent) reduction of body mass index and body weight

SECONDARY OUTCOMES:
(Percent) reduction of: Glucose, cholesterol,LDL, HDL and triglyceride
leptin, adiponectin and ghrelin comparisons and analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD, PhD, Study Director — Chinese Medicine Dep, Taipei Hospital
Locations (1):
- Taipei Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- See also: related research — http://www.nature.com/ijo/journal/v29/n11/abs/0802997a.html
- See also: related research — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=16076989&itool=iconfft&query_hl=2&itool=pubmed_docsum
- See also: related study — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=15976140&itool=iconfft&query_hl=2&itool=pubmed_docsum
- See also: study — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=15738931&itool=iconabstr&query_hl=4&itool=pubmed_docsum